CLINICAL TRIAL: NCT00664183
Title: A Phase 3 Safety and Efficacy Study of Vitreosolve® for Ophthalmic Intravitreal Injection in Retinopathy Subjects
Brief Title: A Safety and Efficacy Study of Vitreosolve® for Non-Proliferative Diabetic Retinopathy Subjects
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: slow enrollment , interim analysis conducted.
Sponsor: Vitreoretinal Technologies, Inc. (Industry)
Responsible Party: Hampar Karageozian, CEO
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PVD-301
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Vitreosolve
- 2 (Experimental)
  Interventions: Drug: Vitreosolve

INTERVENTIONS:
Drug: Vitreosolve — Intravitreal injection

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Vitreosolve in diabetic retinopathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of systemic diabetes (type I or II)
* Subject with a documented history of Non Proliferative Diabetic Retinopathy (NPDR)
* Subjects with no PVD at baseline exam in the study eye.

Exclusion Criteria:

* Subjects with Retinal pathology in the study eye other than (NPDR)
* Subjects with high myopia in the study eye
* Subjects who have monocular vision or contra lateral vision of 20/200 or worse BCVA in the non-study eye.
* Subjects with an aphakic study eye or if pseudophakic, cataract extraction surgery less than 6 months prior to study enrollment
* Subjects that have had either vitrectomy surgery, intravitreal injections, or laser treatments in the study eye.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Ultrasound | 7 Months

SECONDARY OUTCOMES:
Ultrasound, OCT, Safety | 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Kupperman, MD, Principal Investigator — University of California, Irvine; Naresh Mandova, MD, Principal Investigator — University of Colorado, Denver
Locations (17):
- United States (10):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Santa Ana, California
  - Gainesville, Florida
  - Lakeland, Florida
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Asheville, North Carolina
  - McAllen, Texas
  - Silverdale, Washington
- India (7):
  - LVPEI, Bhubhneshwar
  - Sankara Nethralaya, Chennai
  - Aravind, Coimbatore
  - AIIMS, Delhi
  - LVPEI, Hyderabad
  - Aravind, Madurai
  - Aravind, Puducherry